CLINICAL TRIAL: NCT07001423
Title: ChOlecystectomy aFter successFul Endoscopic Common Bile Duct Stone Extraction in Elderly
Acronym: COFFEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Mentula, MD, PhD, Head of Emergency Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8971
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cholecystectomy, Laparoscopic; Choledocholithiasis; Cholelithiasis
MeSH Terms: conditions — Choledocholithiasis; Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecystectomy (Active Comparator): Laparoscopic cholecystectomy is done within 2 weeks after endoscopic removal of common bile duct stones.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Wait-and-see (No Intervention): After endoscopic removal of common bile duct stones, patients are managed non-operatively. During the follow-up cholecystectomy will be available on demand.

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy within 2 weeks after endoscopic removal of common bile duct stone
  Arms: Cholecystectomy

SUMMARY:
The goal of this study is to compare safety and efficacy of laparoscopic cholecystectomy versus wait-and-see policy after endoscopic removal of common bile duct stones in elderly. The primary endpoint is a composite outcome: Death or major postoperative complications or recurrent biliary disease within 1 year after randomization.

DETAILED DESCRIPTION:
Elderly patients with common bile duct stones are asked to participate this randomized trial after successful endoscopic removal of common bile duct stones. The hypothesis of the study is that wait-and-see policy is non-inferior to laparoscopic cholecystectomy. Four hundred patients are randomized 1:1 to either laparoscopic cholecystectomy group or wait-and see group. Cholecystectomy is done on the same admission or within two weeks after randomization. One interim analysis is planned for the trial after 100 randomized patients to assess safety. The trial is terminated if there is a statistically significant difference in primary outcome with p<0.001 (chi-square test) between the study arms.

ELIGIBILITY:
Inclusion Criteria:

* Common bile duct stones cleared after Endoscopic Retrograde Cholangio Pancreatography (ERCP)
* Age >= 80 years or age 75-79 years with a Charlson Comorbidity index >=2
* gallbladder in situ

Exclusion Criteria:

* Acute Cholecystitis
* Biliary Pancreatitis
* Severe or moderately severe post-ERCP pancreatitis
* Chronic pancreatitis
* Bile duct pathology
* Widespread malignancy
* Unable to give consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-03 (Estimated); Primary Completion 2031-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite outcome of death, major complication or recurrent biliary event | From randomization to 1 year
  The primary outcome is a composite outcome including death within 1 year after randomization, the occurrence of major complications within 30 days from surgery and recurrent biliary event requiring hospitalization. within 1 year after randomization. A recurrent biliary event refers to cholecystitis, pancreatitis, cholangitis, or bile duct stones. Major complications were defined as infectious, cardiovascular and pulmonary complications, and surgical complication (Clavien-Dindo grade III or higher)

SECONDARY OUTCOMES:
Number of good days | From randomization to 1 year
  Number of days alive and out of hospital
EQ VAS value | at 30 days, 180 days and 365 days after randomization
  Quality of life is measured using EuroQOL EQ-5D-5L instrument, EQ VAS values are compared. 0 represents the worst health a person can imagine and 100 represents the the best health a person can imagine. EQ-5D-5L dimension responses are reported as a descriptive data
Survival | From randomization to 1 year
  Survival is measured using Kaplan-Meier analysis
Number of patients with major complications | From randomization to 1 year
  Number of patients with major complications defined as infectious, cardiovascular, and pulmonary complications, and surgical complication (Clavien-Dindo grade III or higher)
Number of patients with recurrent biliary event | From randomization to 1 year
  Number of patients with recurrent biliary event (cholecystitis, pancreatitis, cholangitis, or symptomatic bile duct stones)
Composite outcome of death or occurrence of major complications or recurrent biliary event requiring hospitalization | From randomization to 2 years
  The same as primary outcome, but after 2 years follow-up
Number of patients with uncomplicated biliary pain or post cholecystectomy pain | At 30, 180 and 365 days after randomization
  Uncomplicated biliary pain/ post cholecystectomy pain. Specific 5 criteria of biliary pain include : 1. severe pain attacks, 2. lasting 15 to 30 minutes or longer, 3. location in epigastrium or right upper quadrant, 4. pain radiating to the back, 5. a positive pain response to simple analgesics
Healthcare costs | From randomization to 1 year
  Healthcare costs related to bile stones; including laboratory tests, imaging (ultra sound, computer tomography, magnetic resonance imaging), procedures (Endoscopic Retrograde Cholangio Pancreatography (ERCP), laparoscopic cholecystectomy), emergency visits and hospital days.

CONTACTS AND LOCATIONS:
Overall Officials: Panu Mentula, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (12):
- Finland (12):
  - Helsinki University Hospital, Jorvi, Espoo
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Helsinki University Hospital, Meilahti, Helsinki
  - Pohjois-Karjala Central Hospital, Joensuu
  - Keski-Suomi Central Hospital, Jyväskylä
  - Kymenlaakso Central Hospital, Kotka
  - Kuopio University Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kivivuori A, Mattila L, Siiki A, Laukkarinen J, Rantanen T, Ukkonen M. Wait-and-see strategy is justified after ERCP and endoscopic sphincterotomy in elderly patients with common biliary duct stones. J Trauma Acute Care Surg. 2023 Mar 1;94(3):443-447. doi: 10.1097/TA.0000000000003852. Epub 2022 Dec 14. PMID 36524923
- [Background] Costi R, DiMauro D, Mazzeo A, Boselli AS, Contini S, Violi V, Roncoroni L, Sarli L. Routine laparoscopic cholecystectomy after endoscopic sphincterotomy for choledocholithiasis in octogenarians: is it worth the risk? Surg Endosc. 2007 Jan;21(1):41-7. doi: 10.1007/s00464-006-0169-2. Epub 2006 Nov 16. PMID 17111279
- [Background] Boerma D, Rauws EA, Keulemans YC, Janssen IM, Bolwerk CJ, Timmer R, Boerma EJ, Obertop H, Huibregtse K, Gouma DJ. Wait-and-see policy or laparoscopic cholecystectomy after endoscopic sphincterotomy for bile-duct stones: a randomised trial. Lancet. 2002 Sep 7;360(9335):761-5. doi: 10.1016/S0140-6736(02)09896-3. PMID 12241833
- [Background] Bass GA, Gillis AE, Cao Y, Mohseni S; European Society for Trauma and Emergency Surgery (ESTES) Cohort Studies Group. Patients over 65 years with Acute Complicated Calculous Biliary Disease are Treated Differently-Results and Insights from the ESTES Snapshot Audit. World J Surg. 2021 Jul;45(7):2046-2055. doi: 10.1007/s00268-021-06052-0. Epub 2021 Apr 3. PMID 33813631